CLINICAL TRIAL: NCT02058160
Title: A Randomized, 30-week, Active-controlled, Open Label, 2- Treatment Arm, Parallel-group, Multicenter Study Comparing the Efficacy and Safety of the Insulin Glargine/Lixisenatide Fixed Ratio Combination to Insulin Glargine With or Without Metformin in Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Efficacy and Safety of the Insulin Glargine/Lixisenatide Fixed Ratio Combination Versus Insulin Glargine in Patients With Type 2 Diabetes
Acronym: LixiLan-L
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC12405; 2013-003132-79 (EudraCT Number); U1111-1148-4351 (Other: UTN)
Record Dates: First submitted 2014-02-06; First posted 2014-02-07 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) (Experimental): FRC once daily (QD) for 30 weeks. Dose individually adjusted.
  Interventions: Drug: Insulin glargine/lixisenatide (HOE901/AVE0010); Drug: Metformin (Background Drug)
- Insulin glargine (Active Comparator): Insulin glargine 100 U/mL QD for 30 weeks. Dose individually adjusted.
  Interventions: Drug: Insulin glargine (HOE901); Drug: Metformin (Background Drug)

INTERVENTIONS:
Drug: Insulin glargine/lixisenatide (HOE901/AVE0010) — Insulin glargine/lixisenatide FRC was self-administered by subcutaneous (SC) injection within 1 hour before breakfast using one of 2 SoloStar® pen-injectors: Pen A (ratio of 2 Units (U) of insulin glargine U 100:1 mcg of lixisenatide) or Pen B (ratio of 3 U of insulin glargine U 100:1 mcg of lixisenatide). After run-in, the FRC was initiated at a dose of either 20 U/10 mcg with Pen A or 30 U/10 mcg with Pen B, depending on participant's dose of Insulin glargine on the day prior to randomization.
  Dose was adjusted weekly to reach and maintain fasting self-monitored plasma glucose (SMPG) of 80 mg/dL to 100 mg/dL (4.4 mmol/L to 5.6 mmol/L). Pen A was used for administration of doses up to 40 U/20 mcg and Pen B for administration of doses from 30 U/10 mcg up to 60 U/20 mcg.
  Arms: Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC)
Drug: Insulin glargine (HOE901) — Insulin glargine was self-administered QD by SC injection at approximately the same time every day.
  After screening, eligible participants entered 6 week run-in phase during which they were switched (if necessary) to insulin glargine and dose was stabilized. The first dose after randomization was same as the one administered on the day prior to randomization and then dose was adjusted weekly to reach and maintain fasting SMPG of 80 mg/dL to 100 mg/dL (4.4 mmol/L to 5.6 mmol/L).
  Other Names: Lantus
  Arms: Insulin glargine
Drug: Metformin (Background Drug) — Pharmaceutical form: Tablet; Route of administration: Oral administration

SUMMARY:
Primary Objective:

To demonstrate the superiority of the insulin glargine/lixisenatide fixed ratio combination (FRC) to insulin glargine in glycated hemoglobin (HbA1c) change from baseline to Week 30.

Secondary Objective:

To compare the overall efficacy and safety of insulin glargine/lixisenatide FRC to insulin glargine (with or without metformin) over a 30 week treatment period in participants with type 2 diabetes.

DETAILED DESCRIPTION:
Maximum duration of approximately 39 weeks: an up to 8-week screening period, a 30-week randomized treatment period and 3 days post-treatment safety follow up period.

ELIGIBILITY:
Inclusion criteria :

* Type 2 diabetes mellitus diagnosed at least 1 year before the screening visit.
* Treatment with basal insulin for at least 6 months before the screening visit.
* Stable basal insulin regimen (i.e. type of insulin and time/frequency of the injection) for at least 3 months before the screening visit.
* Stable (plus/minus 20 percent) total daily basal insulin dose between 15 and 40 Units/day for at least 2 months prior to the screening visit.
* For participants receiving basal insulin and 1 or 2 oral anti-diabetic drugs (OADs): the OAD dose(s) must be stable during the 3 months before the screening visit. The OADs could be 1 to 2 out of:

  * metformin (more than or equal to 1500 mg/day or maximal tolerated dose),
  * a sulfonylurea,
  * a glinide,
  * a dipeptidyl-peptidase-4 inhibitor,
  * a sodium glucose co-transporter 2 inhibitor,
* Fasting Plasma Glucose (FPG) less than or equal to 180 mg/dL(10.0 mmol/L) at screening visit for participants receiving basal insulin in combination with 2 OADs or with 1 OAD other than metformin; FPG less than or equal to 200 mg/dL (11.1 mmol/L) at screening visit for participants on basal insulin only or basal insulin plus metformin at screening visit.
* Signed written informed consent.

Exclusion criteria:

* Age under legal age of adulthood at screening visit.
* HbA1c at screening visit less than 7.5% or above 10%.
* Pregnancy or lactation, women of childbearing potential with no effective contraceptive method.
* Use of other oral or injectable glucose-lowering agents than stated in the inclusion criteria in a period of 3 months prior to screening.
* Previous use of insulin other than basal insulin eg, prandial or pre-mixed insulin, in the year prior to screening. Note: Short term treatment (≤10 days) due to intercurrent illness is allowed.
* History discontinuation of a previous treatment with Glucagon Like Peptide -1 Receptor Agonists for safety/tolerability or lack of efficacy.
* Participant who had previously participated in any clinical trial with lixisenatide or the insulin glargine/lixisenatide FRC or had previously received lixisenatide.
* Use of weight loss drugs within 3 months prior to screening visit.
* Within the last 6 months prior to screening visit: history of stroke, myocardial infarction, unstable angina, or heart failure requiring hospitalization. Planned coronary, carotid or peripheral artery revascularisation procedures to be performed during the study period.
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy was already performed), chronic pancreatitis, pancreatitis during a previous treatment with incretin therapies, pancreatectomy, stomach/gastric surgery.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (eg, multiple endocrine neoplasia syndromes).
* Uncontrolled or inadequately controlled hypertension (systolic blood pressure above 180 mmHg or diastolic blood pressure above 95 mmHg) at screening visit.
* At screening visit, Body Mass Index (BMI) less than or equal to 20 or above 40 kg/m^2.
* At screening visit amylase and/or lipase more than 3 times the upper limit of the normal (ULN) laboratory range.
* At screening visit alanine aminotransferase (ALT) or alkaline phosphatase (AST) more than 3 ULN.
* At screening visit calcitonin above or equal to 20 pg/mL (5.9 pmol/L).
* Any contraindication to metformin use, according to local labeling, if the participant was taking metformin.
* Participant who had a renal function impairment with creatinine clearance less than 30 mL/min (using the Cockcroft and Gault formula) or end-stage renal disease for participants, not treated with metformin.

Exclusion criteria for randomization:

* HbA1c less than 7% or above 10% .
* Mean fasting SMPG calculated from the self-measurements for 7 days the week before randomization visit was above 140 mg/dL (7.8 mmol/L).
* Average insulin glargine daily dose less than 20 Units or above 50 Units (in the week before randomization visit).
* Amylase and/or lipase more than 3 ULN .

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (236):
- United States (108):
  - Investigational Site Number 840607, Birmingham, Alabama
  - Investigational Site Number 840570, Sun City, Arizona
  - Investigational Site Number 840562, Tempe, Arizona
  - Investigational Site Number 840577, Tucson, Arizona
  - Investigational Site Number 840517, Little Rock, Arkansas
  - Investigational Site Number 840537, Little Rock, Arkansas
  - Investigational Site Number 840568, Bell Gardens, California
  - Investigational Site Number 840550, Chino, California
  - Investigational Site Number 840529, Chula Vista, California
  - Investigational Site Number 840623, Corona, California
  - Investigational Site Number 840566, Fresno, California
  - Investigational Site Number 840552, Greenbrae, California
  - Investigational Site Number 840578, Lancaster, California
  - Investigational Site Number 840626, Los Angeles, California
  - Investigational Site Number 840581, Los Angeles, California
  - Investigational Site Number 840621, Mission Viejo, California
  - Investigational Site Number 840511, Northridge, California
  - Investigational Site Number 840573, Palm Springs, California
  - Investigational Site Number 840559, Port Hueneme, California
  - Investigational Site Number 840536, San Ramon, California
  - Investigational Site Number 840567, Santa Ana, California
  - Investigational Site Number 840569, Tarzana, California
  - Investigational Site Number 840572, West Hills, California
  - Investigational Site Number 840582, Aurora, Colorado
  - Investigational Site Number 840509, Denver, Colorado
  - Investigational Site Number 840549, Wilmington, Delaware
  - Investigational Site Number 840510, Miami, Florida
  - Investigational Site Number 840521, New Port Richey, Florida
  - Investigational Site Number 840602, Ocala, Florida
  - Investigational Site Number 840538, Ocoee, Florida
  - Investigational Site Number 840534, Palm Harbor, Florida
  - Investigational Site Number 840594, Atlanta, Georgia
  - Investigational Site Number 840614, Columbus, Georgia
  - Investigational Site Number 840501, Lawrenceville, Georgia
  - Investigational Site Number 840525, Roswell, Georgia
  - Investigational Site Number 840588, Idaho Falls, Idaho
  - Investigational Site Number 840580, Arlington Heights, Illinois
  - Investigational Site Number 840519, Chicago, Illinois
  - Investigational Site Number 840612, Chicago, Illinois
  - Investigational Site Number 840556, Springfield, Illinois
  - Investigational Site Number 840543, Avon, Indiana
  - Investigational Site Number 840565, Evansville, Indiana
  - Investigational Site Number 840585, Evansville, Indiana
  - Investigational Site Number 840615, Evansville, Indiana
  - Investigational Site Number 840563, Indianapolis, Indiana
  - Investigational Site Number 840507, Indianapolis, Indiana
  - Investigational Site Number 840516, Louisville, Kentucky
  - Investigational Site Number 840595, Lewiston, Maine
  - Investigational Site Number 840520, Baltimore, Maryland
  - Investigational Site Number 840560, Baltimore, Maryland
  - Investigational Site Number 840522, Rockville, Maryland
  - Investigational Site Number 840505, Dearborn, Michigan
  - Investigational Site Number 840575, Flint, Michigan
  - Investigational Site Number 840564, Minneapolis, Minnesota
  - Investigational Site Number 840558, Butte, Montana
  - Investigational Site Number 840506, Omaha, Nebraska
  - Investigational Site Number 840600, Henderson, Nevada
  - Investigational Site Number 840532, Las Vegas, Nevada
  - Investigational Site Number 840599, Las Vegas, Nevada
  - Investigational Site Number 840539, Nashua, New Hampshire
  - Investigational Site Number 840576, Albuquerque, New Mexico
  - Investigational Site Number 840583, Jamaica, New York
  - Investigational Site Number 840531, New Hyde Park, New York
  - Investigational Site Number 840557, Syracuse, New York
  - Investigational Site Number 840541, Durham, North Carolina
  - Investigational Site Number 840604, Greenville, North Carolina
  - Investigational Site Number 840540, Hickory, North Carolina
  - Investigational Site Number 840513, Morehead City, North Carolina
  - Investigational Site Number 840592, Salisbury, North Carolina
  - Investigational Site Number 840535, Wilmington, North Carolina
  - Investigational Site Number 840515, Winston-Salem, North Carolina
  - Investigational Site Number 840579, Columbus, Ohio
  - Investigational Site Number 840524, Dayton, Ohio
  - Investigational Site Number 840503, Maumee, Ohio
  - Investigational Site Number 840618, Eugene, Oregon
  - Investigational Site Number 840610, Philadelphia, Pennsylvania
  - Investigational Site Number 840551, Smithfield, Pennsylvania
  - Investigational Site Number 840584, Tipton, Pennsylvania
  - Investigational Site Number 840622, Charleston, South Carolina
  - Investigational Site Number 840611, Rapid City, South Dakota
  - Investigational Site Number 840605, Amarillo, Texas
  - Investigational Site Number 840553, Austin, Texas
  - Investigational Site Number 840598, Austin, Texas
  - Investigational Site Number 840502, Corpus Christi, Texas
  - Investigational Site Number 840601, Dallas, Texas
  - Investigational Site Number 840586, Dallas, Texas
  - Investigational Site Number 840547, Dallas, Texas
  - Investigational Site Number 840530, Dallas, Texas
  - Investigational Site Number 840545, Dallas, Texas
  - Investigational Site Number 840554, Edinburg, Texas
  - Investigational Site Number 840544, Houston, Texas
  - Investigational Site Number 840514, Hurst, Texas
  - Investigational Site Number 840617, N Richland Hill, Texas
  - Investigational Site Number 840512, Draper, Utah
  - Investigational Site Number 840591, Murray, Utah
  - Investigational Site Number 840526, Ogden, Utah
  - Investigational Site Number 840597, Orem, Utah
  - Investigational Site Number 840590, Salt Lake City, Utah
  - Investigational Site Number 840613, Burlington, Vermont
  - Investigational Site Number 840504, Chesapeake, Virginia
  - Investigational Site Number 840561, Norfolk, Virginia
  - Investigational Site Number 840625, Norfolk, Virginia
  - Investigational Site Number 840606, Richmond, Virginia
  - Investigational Site Number 840608, Salem, Virginia
  - Investigational Site Number 840571, Federal Way, Washington
  - Investigational Site Number 840593, Spokane, Washington
  - Investigational Site Number 840609, Tacoma, Washington
  - Investigational Site Number 840546, Milwaukee, Wisconsin
- Australia (3):
  - Investigational Site Number 036505, Box Hill
  - Investigational Site Number 036501, Heidelberg
  - Investigational Site Number 036504, Parkville
- Canada (11):
  - Investigational Site Number 124504, Beamsville
  - Investigational Site Number 124512, Brampton
  - Investigational Site Number 124502, Guelph
  - Investigational Site Number 124507, Kelowna
  - Investigational Site Number 124505, Montreal
  - Investigational Site Number 124511, Oakville
  - Investigational Site Number 124509, Saint Romuald
  - Investigational Site Number 124503, Toronto
  - Investigational Site Number 124510, Toronto
  - Investigational Site Number 124501, Vancouver
  - Investigational Site Number 124508, Victoria
- Chile (9):
  - Investigational Site Number 152511, Puerto Varas
  - Investigational Site Number 152502, Santiago
  - Investigational Site Number 152501, Santiago
  - Investigational Site Number 152514, Santiago
  - Investigational Site Number 152503, Santiago
  - Investigational Site Number 152507, Santiago
  - Investigational Site Number 152509, Talagante
  - Investigational Site Number 152513, Temuco
  - Investigational Site Number 152504, Viña del Mar
- Czechia (11):
  - Investigational Site Number 203502, Cheb
  - Investigational Site Number 203504, Hranice
  - Investigational Site Number 203507, Krnov
  - Investigational Site Number 203506, Liberec
  - Investigational Site Number 203503, Olomouc
  - Investigational Site Number 203514, Pilsen
  - Investigational Site Number 203515, Pilsen
  - Investigational Site Number 203511, Prague
  - Investigational Site Number 203508, Prague
  - Investigational Site Number 203509, Prague
  - Investigational Site Number 203505, Prostějov
- Denmark (6):
  - Investigational Site Number 208503, Aarhus C
  - Investigational Site Number 208509, Horsens
  - Investigational Site Number 208502, Kolding
  - Investigational Site Number 208501, København NV
  - Investigational Site Number 208505, København S
  - Investigational Site Number 208504, Viborg
- Estonia (3):
  - Investigational Site Number 233502, Pärnu
  - Investigational Site Number 233503, Tallinn
  - Investigational Site Number 233501, Tartu
- Hungary (6):
  - Investigational Site Number 348503, Budapest
  - Investigational Site Number 348501, Budapest
  - Investigational Site Number 348505, Budapest
  - Investigational Site Number 348502, Debrecen
  - Investigational Site Number 348506, Kaposvár
  - Investigational Site Number 348504, Pápa
- Lithuania (5):
  - Investigational Site Number 440501, Kaunas
  - Investigational Site Number 440503, Kaunas
  - Investigational Site Number 440505, Kėdainiai
  - Investigational Site Number 440504, Klaipėda
  - Investigational Site Number 440502, Vilnius
- Mexico (8):
  - Investigational Site Number 484508, Celaya
  - Investigational Site Number 484501, Cuernavaca
  - Investigational Site Number 484503, Guadalajara
  - Investigational Site Number 484504, Guadalajara
  - Investigational Site Number 484506, Guadalajara
  - Investigational Site Number 484509, México
  - Investigational Site Number 484507, Pachuca
  - Investigational Site Number 484505, Puebla City
- Investigational Site Number 528505, Almere Stad, Netherlands
- Poland (7):
  - Investigational Site Number 616502, Bialystok
  - Investigational Site Number 616505, Krakow
  - Investigational Site Number 616506, Krakow
  - Investigational Site Number 616507, Płock
  - Investigational Site Number 616504, Szczecin
  - Investigational Site Number 616503, Warsaw
  - Investigational Site Number 616501, Warsaw
- Romania (11):
  - Investigational Site Number 642507, Brasov
  - Investigational Site Number 642510, Bucharest
  - Investigational Site Number 642508, Bucharest
  - Investigational Site Number 642509, Bucharest
  - Investigational Site Number 642506, Hunedoara
  - Investigational Site Number 642505, Iași
  - Investigational Site Number 642502, Oradea
  - Investigational Site Number 642511, Sibiu
  - Investigational Site Number 642501, Târgu Mureş
  - Investigational Site Number 642504, Timișoara
  - Investigational Site Number 642503, Timișoara
- Russia (13):
  - Investigational Site Number 643511, Arkhangelsk
  - Investigational Site Number 643512, Moscow
  - Investigational Site Number 643508, Penza
  - Investigational Site Number 643501, Saint Petersburg
  - Investigational Site Number 643506, Saint Petersburg
  - Investigational Site Number 643503, Saint Petersburg
  - Investigational Site Number 643504, Saint Petersburg
  - Investigational Site Number 643505, Saint Petersburg
  - Investigational Site Number 643502, Saint Petersburg
  - Investigational Site Number 643513, Samara
  - Investigational Site Number 643507, Saratov
  - Investigational Site Number 643514, Saratov
  - Investigational Site Number 643509, Voronezh
- Slovakia (11):
  - Investigational Site Number 703505, Bratislava
  - Investigational Site Number 703507, Bytča
  - Investigational Site Number 703502, Košice
  - Investigational Site Number 703512, Košice
  - Investigational Site Number 703510, Košice
  - Investigational Site Number 703511, Ľubochňa
  - Investigational Site Number 703508, Moldava nad Bodvou
  - Investigational Site Number 703504, Nové Mesto nad Váhom
  - Investigational Site Number 703509, Nové Zámky
  - Investigational Site Number 703513, Trnava
  - Investigational Site Number 703501, Žilina
- Spain (10):
  - Investigational Site Number 724508, A Coruña
  - Investigational Site Number 724509, Alicante
  - Investigational Site Number 724506, Alzira
  - Investigational Site Number 724504, Barcelona
  - Investigational Site Number 724510, Barcelona
  - Investigational Site Number 724505, Cáceres
  - Investigational Site Number 724503, Ferrol
  - Investigational Site Number 724501, Sabadell
  - Investigational Site Number 724507, Segovia
  - Investigational Site Number 724502, Valencia
- Sweden (6):
  - Investigational Site Number 752501, Ljungby
  - Investigational Site Number 752503, Malmo
  - Investigational Site Number 752504, Rättvik
  - Investigational Site Number 752506, Stenungssund
  - Investigational Site Number 752505, Stockholm
  - Investigational Site Number 752502, Vällingby
- Ukraine (7):
  - Investigational Site Number 804501, Chernivtsi
  - Investigational Site Number 804510, Kyiv
  - Investigational Site Number 804507, Kyiv
  - Investigational Site Number 804511, Kyiv
  - Investigational Site Number 804513, Lviv
  - Investigational Site Number 804502, Vinnytsia
  - Investigational Site Number 804508, Vinnytsia

REFERENCES:
- [Result] Aroda VR, Rosenstock J, Wysham C, Unger J, Bellido D, Gonzalez-Galvez G, Takami A, Guo H, Niemoeller E, Souhami E, Bergenstal RM; LixiLan-L Trial Investigators. Efficacy and Safety of LixiLan, a Titratable Fixed-Ratio Combination of Insulin Glargine Plus Lixisenatide in Type 2 Diabetes Inadequately Controlled on Basal Insulin and Metformin: The LixiLan-L Randomized Trial. Diabetes Care. 2016 Nov;39(11):1972-1980. doi: 10.2337/dc16-1495. Epub 2016 Sep 20. PMID 27650977
- [Derived] Tabak AG, Anderson J, Aschner P, Liu M, Saremi A, Stella P, Tinahones FJ, Wysham C, Meier JJ. Efficacy and Safety of iGlarLixi, Fixed-Ratio Combination of Insulin Glargine and Lixisenatide, Compared with Basal-Bolus Regimen in Patients with Type 2 Diabetes: Propensity Score Matched Analysis. Diabetes Ther. 2020 Jan;11(1):305-318. doi: 10.1007/s13300-019-00735-7. Epub 2019 Dec 17. PMID 31848983
- [Derived] Blonde L, Bailey TS, Chao J, Dex TA, Frias JP, Meneghini LF, Roberts M, Aroda VR. Clinical Characteristics and Glycemic Outcomes of Patients with Type 2 Diabetes Requiring Maximum Dose Insulin Glargine/Lixisenatide Fixed-Ratio Combination or Insulin Glargine in the LixiLan-L Trial. Adv Ther. 2019 Sep;36(9):2310-2326. doi: 10.1007/s12325-019-01033-1. Epub 2019 Jul 29. PMID 31359368
- [Derived] Dailey G, Bajaj HS, Dex T, Groleau M, Stager W, Vinik A. Post hoc efficacy and safety analysis of insulin glargine/lixisenatide fixed- ratio combination in North American patients compared with the rest of world. BMJ Open Diabetes Res Care. 2019 Mar 21;7(1):e000581. doi: 10.1136/bmjdrc-2018-000581. eCollection 2019. PMID 31114694
- [Derived] Schmider W, Belder R, Lee M, Niemoeller E, Souhami E, Frias JP. Impact of dose capping in insulin glargine/lixisenatide fixed-ratio combination trials in patients with type 2 diabetes. Curr Med Res Opin. 2019 Jun;35(6):1081-1089. doi: 10.1080/03007995.2018.1558852. Epub 2019 Jan 11. PMID 30550345
- [Derived] Zisman A, Dex T, Roberts M, Saremi A, Chao J, Aroda VR. Bedtime-to-Morning Glucose Difference and iGlarLixi in Type 2 Diabetes: Post Hoc Analysis of LixiLan-L. Diabetes Ther. 2018 Oct;9(5):2155-2162. doi: 10.1007/s13300-018-0507-0. Epub 2018 Sep 14. PMID 30218434
- [Derived] Rosenstock J, Handelsman Y, Vidal J, Ampudia Blasco FJ, Giorgino F, Liu M, Perfetti R, Meier JJ. Propensity-score-matched comparative analyses of simultaneously administered fixed-ratio insulin glargine 100 U and lixisenatide (iGlarLixi) vs sequential administration of insulin glargine and lixisenatide in uncontrolled type 2 diabetes. Diabetes Obes Metab. 2018 Dec;20(12):2821-2829. doi: 10.1111/dom.13462. Epub 2018 Aug 13. PMID 29974618
- [Derived] Trujillo JM, Roberts M, Dex T, Chao J, White J, LaSalle J. Low incidence of gastrointestinal adverse events over time with a fixed-ratio combination of insulin glargine and lixisenatide versus lixisenatide alone. Diabetes Obes Metab. 2018 Nov;20(11):2690-2694. doi: 10.1111/dom.13444. Epub 2018 Aug 21. PMID 29923298
- [Derived] Niemoeller E, Souhami E, Wu Y, Jensen KH. iGlarLixi Reduces Glycated Hemoglobin to a Greater Extent Than Basal Insulin Regardless of Levels at Screening: Post Hoc Analysis of LixiLan-L. Diabetes Ther. 2018 Feb;9(1):373-382. doi: 10.1007/s13300-017-0336-6. Epub 2017 Nov 16. PMID 29143919
- [Derived] Wysham C, Bonadonna RC, Aroda VR, Puig Domingo M, Kapitza C, Stager W, Yu C, Niemoeller E, Souhami E, Bergenstal RM; LixiLan-L trial investigators. Consistent findings in glycaemic control, body weight and hypoglycaemia with iGlarLixi (insulin glargine/lixisenatide titratable fixed-ratio combination) vs insulin glargine across baseline HbA1c, BMI and diabetes duration categories in the LixiLan-L trial. Diabetes Obes Metab. 2017 Oct;19(10):1408-1415. doi: 10.1111/dom.12961. Epub 2017 Jun 8. PMID 28386990

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 236 centers in 18 countries. A total of 1930 participants were screened between January 27, 2014 and October 15, 2014. 912 participants were not eligible for run-in-phase mainly due to glycated hemoglobin (HbA1c) value being out of the protocol defined range.
Pre-assignment Details: After screening phase, 1018 participants entered 6 week run-in phase during which participants were switched (if necessary) to insulin glargine and dose was titrated/stabilized, any oral anti-diabetic drugs (OAD) other than metformin were stopped. 282 participants were run-in failures and 736 were randomized in 1:1(FRC:insulin glargine arms) ratio.
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC): FRC injected subcutaneously once daily (QD) for 30 weeks. Dose individually adjusted.
- Insulin Glargine: Insulin glargine 100 U/mL injected subcutaneously QD for 30 weeks. Dose individually adjusted.
Period: Overall Study
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination (FRC) | Insulin Glargine
Started | 367 | 369
Treated | 365 | 365
Completed | 336 | 355
Not Completed | 31 | 14
Not completed — Randomized but not treated | 2 | 4
Not completed — Poor compliance to protocol | 4 | 1
Not completed — Adverse Event | 12 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other than specified above | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination: FRC injected subcutaneously QD for 30 weeks. Dose individually adjusted.
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Total
Number analyzed (Participants) | 367 | 369 | 736
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (9.4) | 60.3 (8.7) | 60.0 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 190 | 392
  Male | 165 | 179 | 344
Race [Count of Participants; unit: Participants]
  Caucasian | 337 | 338 | 675
  Black | 17 | 21 | 38
  Asian/Oriental | 12 | 8 | 20
  Other | 1 | 2 | 3
Ethnicity [Count of Participants; unit: Participants]
  Hispanic | 66 | 66 | 132
  Not Hispanic | 301 | 303 | 604
OAD Use [Count of Participants; unit: Participants]
  Yes | 349 | 350 | 699
  No | 18 | 19 | 37
OAD Use at Screening by Class [Count of Participants; unit: Participants]
  Metformin | 170 | 190 | 360
  Sulfonylurea | 16 | 14 | 30
  Sodium glucose co-transporter 2 (SGLT-2) inhibitor | 0 | 1 | 1
  Dipeptidyl-peptidase 4 (DPP-4) inhibitor | 2 | 4 | 6
  Glinide | 1 | 1 | 2
  Metformin + Sulfonylurea | 137 | 118 | 255
  Metformin + DPP-4 inhibitor | 20 | 18 | 38
  Metfomrin + Glinide | 2 | 3 | 5
  Sulfonylurea + DPP-4 inhibitor | 1 | 1 | 2
  None | 18 | 19 | 37
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.33 (4.25) | 30.96 (4.15) | 31.14 (4.20)
Duration of Diabetes [Mean (Standard Deviation); unit: years] — Population: Only participants with available data for this baseline measure were included in the analysis.
  years
    number analyzed (Participants) | 367 | 368 | 735
    (all) | 12.02 (6.64) | 12.13 (6.85) | 12.08 (6.74)
Daily Dose of Metformin [Mean (Standard Deviation); unit: mg] — Population: Only participants with available data for this baseline measure were included in the analysis.
  mg
    number analyzed (Participants) | 329 | 329 | 658
    (all) | 2082.8 (499.2) | 2042.0 (455.9) | 2062.4 (478.1)
Screening Glycated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.51 (0.65) | 8.54 (0.67) | 8.53 (0.66)
Baseline HbA1c [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.07 (0.68) | 8.08 (0.73) | 8.08 (0.71)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 7.34 (1.95) | 7.36 (2.12) | 7.35 (2.04)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Hemoglobin (HbA1c) From Baseline to Week 30
Description: Change in HbA1c was calculated by subtracting baseline value from Week 30 value.
Time Frame: Baseline, Week 30
Population: Modified intent-to-treat (mITT) population: all randomized participants who had both baseline and at least one post-baseline efficacy assessment. Here, number of participants analyzed = participants with baseline and at least one post-baseline HbA1c assessment during study period.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 364 | 364
percentage of HbA1c | -1.13 (0.057) | -0.62 (0.055)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Analysis was performed using Mixed-effect model with repeated measures (MMRM) with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of metformin use at screening, visits, treatment-by-visit interaction and country as fixed effects and baseline HbA1c value-by-visit interaction as covariates. A hierarchical testing procedure was used to control type I error and handle multiple endpoint analyses; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; Least square (LS) mean difference = -0.52, 95% CI 2-sided [-0.633 to -0.397], Standard Error of Mean 0.06 — Insulin Glargine/Lixisenatide FRC vs Insulin Glargine

2. Secondary Outcome: Percentage of Participants With HbA1c <7.0% or ≤6.5% at Week 30
Time Frame: Week 30
Population: mITT population. Participants with no value for HbA1c at Week 30 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 366 | 365
percentage of participants
  HbA1c <7.0% | 54.9 | 29.6
  HbA1c ≤ 6.5% | 33.9 | 14.2
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; HbA1c <7.0%: Insulin Glargine/Lixisenatide FRC vs Insulin Glargine. Analysis was performed using Cochran-Mantel-Haenszel method stratified on randomization strata of Week -1 HbA1c (<8.0%, ≥8.0%) and randomization strata of metformin use at screening. This analysis was out of testing order; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Difference in percentage = 25.52, 95% CI 2-sided [18.94 to 32.10] — HbA1c <7.0%: Insulin Glargine/Lixisenatide FRC vs Insulin Glargine
Statistical Analysis 2: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; HbA1c ≤6.5%: Insulin Glargine/Lixisenatide FRC vs Insulin Glargine. Analysis was performed using Cochran-Mantel-Haenszel method stratified on randomization strata of Week -1 HbA1c (<8.0%, ≥8.0%) and randomization strata of metformin use at screening. This analysis was out of testing order; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentage = 19.76, 95% CI 2-sided [13.90 to 25.62] — HbA1c ≤6.5%: Insulin Glargine/Lixisenatide FRC vs Insulin Glargine

3. Secondary Outcome: Change in 2-hour Plasma Blood Glucose Excursion From Baseline to Week 30
Description: Plasma glucose excursion = 2-hour postprandial glucose (PPG) minus plasma glucose value obtained 30 minutes prior to the start of the meal and before investigational medicinal product (IMP) administration, if IMP was injected before breakfast. Change in plasma glucose excursions was calculated by subtracting baseline value from Week 30 value.
Time Frame: Baseline, Week 30
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline plasma glucose excursion assessment during study period. Missing data was imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 329 | 336
mmol/L | -3.9 (0.285) | -0.47 (0.274)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using analysis of covariance (ANCOVA) model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of metformin use at screening and country as fixed effects and baseline 2-hour plasma glucose excursion value as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -3.43, 95% CI 2-sided [-3.925 to -2.939], Standard Error of Mean 0.251 — Insulin Glargine/Lixisenatide FRC vs Insulin Glargine

4. Secondary Outcome: Change in Body Weight From Baseline to Week 30
Description: Change in body weight was calculated by subtracting baseline value from Week 30 value.
Time Frame: Baseline, Week 30
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline body weight assessment during study period.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 365 | 365
kg | -0.67 (0.181) | 0.7 (0.178)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using MMRM model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of metformin use at screening, scheduled visits, treatment-by-visit interaction and country as fixed effects and baseline body weight value-by-visit interaction as covariates; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -1.37, 95% CI 2-sided [-1.808 to -0.93], Standard Error of Mean 0.224 — Insulin Glargine/Lixisenatide FRC vs Insulin Glargine

5. Secondary Outcome: Mean Change in 7-point Self-monitored Plasma Glucose (SMPG) Profile From Baseline to Week 30
Description: Participants recorded a 7-point plasma glucose profile measured before and 2-hours after each meal and at bedtime, two times in a week before baseline, before visit Week 12 and before visit Week 30 and the average value across the profiles performed in the week before a visit for the 7 time points was calculated. Change in average 7 point SMPG was calculated by subtracting baseline value from Week 30 value. The analysis included all scheduled measurements obtained during the study. The missing data was handled by mixed effect model with repeated measures (MMRM) approach.
Time Frame: Baseline, Week 30
Population: mITT population. Here, number of participants analyzed= participants with baseline and at least one post-baseline 7-point SMPG assessment during study period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 323 | 320
mmol/L | -1.5 (0.137) | -0.6 (0.13)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using MMRM model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of metformin use at screening, scheduled visits, treatment-by-visit interaction and country as fixed effects and baseline average SMPG value-by-visit interaction as covariates; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -0.9, 95% CI 2-sided [-1.154 to -0.64], Standard Error of Mean 0.131 — Insulin Glargine/Lixisenatide FRC vs Insulin Glargine

6. Secondary Outcome: Percentage of Participants Reaching HbA1c <7.0% With No Body Weight Gain at Week 30
Time Frame: Week 30
Population: mITT population. Participants without HbA1c and/or body weight value at Week 30 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 366 | 365
percentage of participants | 34.2 | 13.4
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using Cochran-Mantel-Haenszel method stratified on randomization strata of Week -1 HbA1c (<8.0%, ≥8.0%) and randomization strata of metformin use at screening; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentage = 20.82, 95% CI 2-sided [14.98 to 26.66] — Insulin Glargine/Lixisenatide FRC vs Insulin Glargine

7. Secondary Outcome: Change in Daily Insulin Glargine Dose From Baseline to Week 30
Time Frame: Baseline, Week 30
Population: mITT population. The analysis included scheduled measurements obtained up to the date of last injection of IMP. Here, number of participants analyzed= participants with insulin glargine dose assessment during study period.
Measure: Least Squares Mean (Standard Error); unit: Units (U)
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 364 | 365
Units (U) | 10.64 (0.601) | 10.89 (0.587)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the hierarchical testing procedure (continued only if previous endpoints were statistically significant). Analysis was performed using MMRM model with treatment groups, randomization strata of Week -1 HbA1c (<8.0, ≥8.0%), randomization strata of metformin use at screening, scheduled visits, treatment-by-visit interaction and country as fixed effects and baseline daily insulin glargine dose-by-visit interaction as a covariate; Test type: Superiority or Other; p = 0.7362, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -0.26, 95% CI 2-sided [-1.762 to 1.246], Standard Error of Mean 0.766 — Insulin Glargine/Lixisenatide FRC vs Insulin Glargine

8. Secondary Outcome: Percentage of Participants Reaching HbA1c <7.0% With No Body Weight Gain at Week 30 and No Documented Symptomatic Hypoglycemia (Plasma Glucose [PG] ≤ 70 mg/dL [3.9 mmol/L]) During 30-Week Treatment Period
Description: Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of ≤70 mg/dL (3.9 mmol/L).
Time Frame: Baseline up to Week 30
Population: mITT population. Participants without HbA1c and/or body weight value at Week 30 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 366 | 365
percentage of participants | 19.9 | 9.0

9. Secondary Outcome: Change in FPG From Baseline to Week 30
Description: Change in FPG was calculated by subtracting baseline value from Week 30 value.
Time Frame: Baseline, Week 30
Population: mITT population. Here, number of participants analyzed= participants with baseline and at least one post-baseline FPG assessment during study period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 364 | 364
mmol/L | -0.35 (0.142) | -0.46 (0.138)

10. Secondary Outcome: Change in 2-hour PPG From Baseline to Week 30
Description: Change in PPG was calculated by subtracting baseline value from Week 30 value.
Time Frame: Baseline, Week 30
Population: mITT population. Here, number of participants analyzed= participants with baseline and at least one post-baseline PPG assessment during study period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 332 | 340
mmol/L | -4.72 (0.322) | -1.39 (0.31)

11. Secondary Outcome: Percentage of Participants Reaching HbA1c <7.0% With No Documented Symptomatic Hypoglycemia (PG ≤ 70 mg/dL [3.9 mmol/L]) During 30-Week Treatment Period
Description: as for outcome 8
Time Frame: Baseline up to Week 30
Population: mITT population. Participants with no value for HbA1c at Week 30 were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 366 | 365
percentage of participants | 31.7 | 18.6

12. Secondary Outcome: Percentage of Participants Requiring Rescue Therapy During 30-Week Treatment Period
Description: Routine fasting SMPG and central laboratory FPG (and HbA1c after Week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after Week 12) were performed. Threshold values - from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 30: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >8%.
Time Frame: Baseline up to Week 30
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 366 | 365
percentage of participants | 2.7 | 6

13. Secondary Outcome: Number of Documented Symptomatic Hypoglycemia Events Per Subject-Year
Description: as for outcome 8
Time Frame: First dose of study drug up to 1 day after the last dose administration (median treatment exposure 211 days [FRC], 210 days [Insulin glargine])
Population: Analysis was performed on safety population defined as all randomized participants who received at least one dose of IMP regardless of the amount of treatment administered.
Measure: Number; unit: events per subject-year
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 365 | 365
events per subject-year | 3.03 | 4.22

14. Secondary Outcome: Percentage of Participants With Documented Symptomatic Hypoglycemia
Description: as for outcome 8
Time Frame: as for outcome 13
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 365 | 365
percentage of participants | 40 | 42.5

15. Secondary Outcome: Percentage of Participants With Severe Symptomatic Hypoglycemia
Description: Severe symptomatic hypoglycemia was an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Plasma glucose measurements might not had been available during such an event, but neurological recovery attributable to the restoration of plasma glucose to normal was considered sufficient evidence that the event had been induced by a low plasma glucose concentration. Severe symptomatic hypoglycemia included all episodes in which neurological impairment was severe enough to prevent self-treatment, and which were thus thought to place participants at risk for injury to themselves or others.
Time Frame: as for outcome 13
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 365 | 365
percentage of participants | 1.1 | 0.3

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 30) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent that is AEs that developed/worsened during 'on-emergent period' (time from first injection of open-label IMP up to 3 days after the last injection of IMP). Analysis was performed on safety population.
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination: FRC injected subcutaneously QD for 30 weeks. Dose individually adjusted (median exposure: 211 days).
- Insulin Glargine: Insulin glargine 100 U/mL injected subcutaneously QD for 30 weeks. Dose individually adjusted (median exposure: 210 days).
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 20/365 | 18/365
Other Adverse Events (participants affected / at risk) | 81/365 | 42/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glargine/Lixisenatide Fixed Ratio Combination (N=365) | Insulin Glargine (N=365)
Pneumonia (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 | 0
Hypoglycaemic seizure (Nervous system disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 2 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Scar (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glargine/Lixisenatide Fixed Ratio Combination (N=365) | Insulin Glargine (N=365)
Nasopharyngitis (Infections and infestations) | 32 | 32
Headache (Nervous system disorders) | 21 | 10
Nausea (Gastrointestinal disorders) | 38 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.